CLINICAL TRIAL: NCT04089631
Title: Circulating Tumour DNA Based Decision for Adjuvant Treatment in Colon Cancer Stage II Evaluation (CIRCULATE) AIO-KRK-0217
Brief Title: Circulating Tumour DNA Based Decision for Adjuvant Treatment in Colon Cancer Stage II Evaluation
Acronym: CIRCULATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUD-CIRC01-071; 2018-003691-12 (EudraCT Number); 01KG1817 (Other Grant/Funding Number: German Federal Ministry for Education and Research (BMBF)); AIO-KRK-0217 (Other: Arbeitsgemeinschaft Internistische Onkologie)
Record Dates: First submitted 2019-09-09; First posted 2019-09-13 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Colon Cancer Stage II
Keywords: circulating tumour DNA; ctDNA; adjuvant chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Experimental): Capecitabine mono or Capecitabine/Oxaliplatin as investigator choice:
  Patients who are positive for postoperative ctDNA (ctDNApos) and not microsatellite instable are randomized (2:1) to adjuvant chemotherapy with capecitabine or to follow up.
  Capecitabine 2 x 1250 mg/m^2, oral (d1-14), repeated at day 22 (- 2 ... + 6 days). Patients with a GFR between 30 and 50 ml/min start with capecitabine dose of 2 x 1000 mg/m^2. Treatment duration: 8 cycles (approx. 6 months)
  Capecitabine, if combined with Oxaliplatin (investigator choice):
  If the investigation decides to add oxaliplatin, the following schedule should be used:
  [Oxaliplatin 130 mg/m^2 i.v. (2 hours on d1)] Capecitabine 2 x 1000 mg/m^2, oral (d1-14), repeated at day 22 (- 2 ... + 6 days) Treatment duration: 4 or 8 cycles (approx. 3 or 6 months)
  Interventions: Drug: Capecitabine
- Follow-up (No Intervention): Patients negative for postoperative ctDNA (ctDNAneg) are randomized (1:4) to follow-up within CIRCULATE or to routine follow up outside the Trial protocol.

INTERVENTIONS:
Drug: Capecitabine — 6 months capecitabine, in combination with oxaliplatin 3 to 6 months capecitabine
  Other Names: Xeloda
  Arms: Chemotherapy

SUMMARY:
The CIRCULATE study evaluates the adjuvant therapy in patients with colon cancer UICC stage II. The primary aim of the study is to compare the disease free survival in patients who are positive for postoperative circulating tumour DNA with vs. without capecitabine.

DETAILED DESCRIPTION:
CIRCULATE is an investigator-initiated, multicentre, prospective, randomised, controlled trial.

Screening phase:

Patients with colon cancer (or rectal cancer, if a radiation is not indicated i.e. due to the tumour localisation) are postoperatively screened for this trial.

For this purpose, they sign an informed consent for screening. The formalin fixed paraffin embedded (FFPE) tumour block is shipped to one of the central pathological laboratories and is analysed for microsatellite instability and by panel analysis for frequent mutations in the colorectal cancer. A plasma sample is sent in parallel to the central laboratory for ctDNA. The screening is preferably performed before the patient is discharged from the surgical department and at the latest 5 weeks after resection to allow sufficient time for the analysis.

The patient- specific tumour mutations known from the panel analysis are measure in the patients plasma by ultra deep sequencing. The results of the analysis - positive for circulating tumour DNA (ctDNApos) or negative for circulating tumour DNA (ctDNAneg) - is not communicated to the patient or the investigator.

Randomised phase:

Four to eight weeks after resection, the patient presents at an investigator that is experienced with chemotherapy (i.e. Medical Oncologist) and consent for the randomised part of the study with a second informed consent form. If this baseline visit confirms that there are not contraindications to chemotherapy and if no other exclusion criteria exist, the patient is randomised:

* ctDNApos patients are randomised (2:1) in "chemotherapy" (with capecitabine) or "follow-up",
* ctDNAneg patients are randomised (1:4) in "follow-up" or "off study" which means that the follow-up will be organised within the routine clinical practice.

The result of the ctDNA will not be communicated to the patients and investigators, so that patients in the arm "follow-up" remain blinded to the ctDNA result. Due to the randomisation ratio, the prognosis of these patients is similar to those in stage II without any ctDNA analysis and differs only slightly from patients not enrolled into a clinical trial.

Patients in the arm "chemotherapy" receive adjuvant therapy with 6 months capecitabine. The investigator can decide to add oxaliplatin and to shorten the adjuvant chemotherapy to 3 months if oxaliplatin is added.

Patients in the arms "chemotherapy" and "follow-up" are followed with the same methods and time point within the study.

Patients in the arm "off study" are recommended to be follow up according to the guidelines for stage II in the routine practice.

ELIGIBILITY:
Inclusion criteria for screening phase:

1. Resected colon cancer stage II, OR Resected rectal cancer stage II, if there was no indication for radiotherapy (i.e. due to the localisation in the upper third of the rectum ), so that the treatment follows the recommendations for colon cancer. Patients, in whom the tumour stage is not yet know, can be enrolled into the screening.
2. Signed informed consent for the screening Phase

Inclusion criteria for the randomised phase:

1. Resected colon cancer stage II, OR resected rectal cancer stage II, if there was no indication for radiotherapy (i.e. due to the localisation in the upper third of the rectum), so that the treatment follows the recommendations for colon cancer.
2. Known microsatellite or mismatch repair status
3. Confirmation, that the ctDNA result is available
4. Signed second informed consent (for the randomised phase)

Exclusion criteria for Screening:

1. Patients with known microsatellite instability (MSI-H) or mismatch repair deficiency (dMMR)
2. Known clinical high risk situation if it is regarded as certain indication for an adjuvant chemotherapy
3. Patients, who have an obvious contra-indication for adjuvant chemotherapy (i.e. due to the performance status, comorbidity, active second cancer or age). It should be considered that patients with an age of more than 75 years frequently not fulfil criteria for adjuvant chemotherapy.
4. R1- or R2-status (patients with [still] unknown R-status can be screened)
5. Patients, in whom the randomisation or chemotherapy is unfeasible due to logistic reasons (travel distance, compliance)
6. Age < 18 years
7. Pregnant or breast feeding patients

Exclusion criteria for randomised phase:

1. Patients with microsatellite instability (MSI-H) or mismatch repair deficiency (dMMR)
2. Known clinical high risk situation if it is regarded as certain indication for an adjuvant chemotherapy
3. R1- or R2- status, or unknown R- status (Rx)
4. Number of investigated lymph nodes < 10
5. WHO performance status ≥ 2
6. Colon or rectal cancer with UICC stage III or IV
7. Second cancer, except

   1. simultaneous or metachronous colon or rectal cancer with UICC stage ≤ I,
   2. curatively treated basal cell carcinoma or squamous cell carcinoma of the skin and in-situ cervical carcinoma
   3. tumours with a disease free survival of more than five years
8. Contra indications for chemotherapy, especially:

   1. Leukocytes < 3,0 Gpt/l
   2. Neutrophil granulocytes < 1,5 Gpt/l
   3. Thrombocytes < 100 Gpt/l
   4. alanine aminotransferase (ALAT) or (aspartate aminotransferase) ASAT > 3x ULN
   5. Creatinine clearance (calculated according Cockcroft-Gault) < 30 ml/min
9. Comorbidities relevantly interfering with the prognosis of the patients, i.e.:

   1. heart insufficiency NYHA III/IV
   2. relevant coronary heart disease,
   3. Diabetes mellitus with late sequelae
10. Organ, stem cell or bone marrow transplantation
11. Known hypersensitivity to capecitabine In case of known hypersensitivity to oxaliplatin, the patients can participate, but not receive oxaliplatin
12. Medication with brivudine, sorivudine or analogues in the last four weeks before planned treatment start
13. Known dihydropyrimidine dehydrogenase (DPD)-deficiency
14. Acute infections
15. Known HIV- infections, known active hepatitis B or C-infection
16. Participation at another interventional study for medical treatment during the last four weeks before randomisation
17. Neoadjuvant therapy before resection
18. Patients, in whom the randomisation or chemotherapy is unfeasible due to logistic reasons (travel distance, compliance)
19. Age < 18 years
20. Pregnant or breast feeding patients
21. Women of childbearing potential and men with partner with childbearing potential who are not willing to take appropriate precautions to avoid pregnancy with a highly effective method in case they are randomised to "chemotherapy"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4812 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Disease free Survival (DFS) | for the primary endpoint after 154 events (approx. 60 months after study start)
  Disease free survival of ctDNA positive patients randomised to "chemotherapy" vs. "follow-up", measured from randomisation to any recurrence, metastasis, second colorectal or non colorectal cancer and death from any cause. The primary endpoint will be tested in all randomised ctDNA positive patients and be evaluated by a stratified log rank test.
  Interims analysis after 93 events (approx. 38 months after study start), final analysis for the primary endpoint after 154 events (approx. 60 months after study start).

SECONDARY OUTCOMES:
Overall survival in ctDNApos patients with adjuvant therapy vs follow-up | 5 years
  Overall survival in ctDNApos patients with adjuvant therapy vs follow-up, measured from randomisation to death from any cause, in all randomised ctDNA positive patients and be evaluated by a stratified log rank test.
Disease free survival in ctDNAneg patients randomised to follow up | 3 years
  Disease free survival in ctDNAneg patients randomised to follow up (rate of patients disease free and alive 3 years after randomisation according to Kaplan-Meier estimation with 95% CI, intention-to-treat analysis). Any recurrence, metastasis, second colorectal or non-colorectal cancer and death from any cause is regarded as event (rate of patients disease free and alive 3 years after randomisation according to Kaplan-Meier estimation with 95% CI, intention-to-treat analysis). Any recurrence, metastasis, second colorectal or non- colorectal cancer and death from any cause is regarded as event
Overall survival in ctDNAneg patients randomised to "follow up" | 5 years
  Overall survival in ctDNAneg patients randomised to "follow up" (rate of patients alive after 5 years after randomisation according to Kaplan-Meier estimation with 95% CI)
Disease free and overall survival of ctDNApos vs. ctDNAneg patients randomized to "follow-up" | 3 years and 5 years
  Disease free and overall survival of ctDNApos vs. ctDNAneg patients randomized to "follow-up" (measured from randomisation to the event in an intention-to-treat analysis by stratified log rank test). Any recurrence, metastasis, second colorectal or non-colorectal cancer and death from any cause are regarded as event for DFS. Death of any cause will be regarded as event for overall survival.
Site of metastases | 5 years
  Site of metastases (lymph node vs. peritoneal/local recurrence vs other) in ctDNApos vs. ctDNAneg patients who have a recurrence / metastases
Frequency of adverse events from start of chemotherapy until 30 days after chemotherapy | 5 years
  Frequency of adverse events from start of chemotherapy until 30 days after chemotherapy (descriptive analysis for patients randomised to "chemotherapy" who have received at least one dose of chemotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Folprecht, Prof., Principal Investigator — University hospital "Carl Gustav Carus" Dresden
Locations (1):
- Universitaetsklinikum Carl Gustav Carus, Medizinische Klinik, Dresden, Saxony, Germany